CLINICAL TRIAL: NCT05875558
Title: Lipiodol Combined With Microspheres TACE for Unresectable HCC
Brief Title: M-TACE Treatment for Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Zhiping Yan, Director, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-ZS-IR-06
Record Dates: First submitted 2023-05-11; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- M-TACE (Experimental)
  Interventions: Procedure: M-TACE

INTERVENTIONS:
Procedure: M-TACE — Lipiodol combined with microspheres

SUMMARY:
This study aims to investigate the safety and efficacy of transarterial chenmoembolization（TACE） combined with microspheres for unresectable hepatocellular carcinoma(HCC).

ELIGIBILITY:
Inclusion Criteria:

1. 18≤Age<80 on day of signing informed consent.
2. Have histologically confirmed diagnosis or radiological diagnosis of HCC with at least one >3cm targeted lesion.
3. Have Barcelona Clinic Liver Cancer (BCLC) Stage C disease or BCLC Stage B disease, BCLC stage A disease but refuse a surgical or ablation therapy.
4. Have a Child-Pugh Class A/B（<7） liver score.
5. Have a performance status of 0 or 1 using the ECOG.
6. Have a predicted life expectancy of greater than 3 months.

Exclusion Criteria:

1. The targeted lesions have received TACE or other locoregional therapy within 3 months.
2. Tumor burden over 70% of the liver volume.
3. Lesions can not be measured by mRECIST.
4. Has a diagnosed additional malignancy.
5. Patients with Hb<9.0g/dL, WBC<1.0×10^9/L， TB>3mg/dL，ALT/AST>5 UL, ALB<2.8g/dL， INR>2.3, Cr >2mg/mL or CCr<30mL/min.
6. Severe heart, lung or cerebral disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 month after first mTACE
  Objective response rate according to the mRECIST
ORR | 3 months after first mTACE
  Objective response rate according to the mRECIST

SECONDARY OUTCOMES:
OS | 1 year
  Overall survival
OS | 3 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Interventional Radiology, Zhongshan Hospital, Fudan University., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No